CLINICAL TRIAL: NCT00003365
Title: The Effect of Plant Phenolic Compounds on Human Colon Epithelial Cells
Brief Title: Sulindac and Plant Compounds in Preventing Colon Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study completed
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Stephen Shiff, UMDNJ
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000066350; P30CA016056 (NIH); RUH-SSH-190-0600; RUH-SSH-190-0698; NCI-V98-1425
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Colorectal Cancer
Keywords: colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Curcumin; Rutin; Quercetin; Sulindac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: curcumin
Dietary Supplement: rutin
Drug: quercetin
Drug: sulindac

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of sulindac may be an effective way to prevent colon cancer. Eating a diet rich in fruits and vegetables appears to reduce the risk of some types of cancer. Curcumin, rutin, and quercetin are compounds found in plants that may prevent the development of colon cancer.

PURPOSE: Randomized clinical trial to study the effectiveness of sulindac, curcumin, rutin, and quercetin in preventing colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response of the colonic epithelium in normal volunteers at average or above average risk of colon cancer, when given short term treatment with plant phenolics such as curcumin, rutin, and quercetin.
* Compare the colonic mucosal response to the plant phenolics with their response to sulindac in order to evaluate whether they share common mechanisms for colon cancer chemoprevention.
* Determine the lowest optimal dose for each of the three plant phenolics that is effective in modulating biomarkers of colon epithelial cell turnover and, therefore, potentially inhibiting colon cancer development.
* Assess the response of the colonic epithelium to curcumin in volunteers at average risk of colon cancer development.

OUTLINE: This is a randomized, controlled, two part, single institution study. Patients in Part B are randomized by gender.

All patients undergo flexible sigmoidoscopic exam.

* Part A: Patients, in cohorts of 5-10, receive one of the following five treatments in addition to the control diet: nothing (arm I), oral sulindac twice a day (arm II), oral rutin at 1 of 3 doses twice a day (arms III, IV, and V), oral quercetin at 1 of 3 doses twice a day (arms V, VI, and VII), or at 1 of 3 doses oral curcumin twice a day (arms VIII, IX, and X). Patients are first randomized to the highest doses of rutin, quercetin, and curcumin and then lower doses may be given in order to determine the minimally effective dose. Treatment is continued for 6-10 weeks.
* Part B: Patients are randomized to receive the control diet only (arm I) or the control diet plus oral curcumin twice a day (arm II) for 6-10 weeks.

Patients are followed every 2 weeks.

PROJECTED ACCRUAL: There will be 130 patients (110 in Part A and 20 in Part B) accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Individuals at average risk (Parts A and B) or above average risk (Part A only) for development of colon cancer

  * Average risk individuals defined as:

    * No history of colon adenomas
    * No strong family history of colon polyps or cancer
  * Above average risk individuals defined as:

    * History of one or more sporadic adenomatous polyps at least 0.5 cm in size (either tubular, tubulovillous, or villous adenomas)
    * Have had polypectomy or refused this procedure
    * No significant family history of adenomatous polyps, colon cancer, or hereditary nonpolyposis colorectal cancer or other hereditary colon cancer syndrome
    * Polyps should not have had a focus of adenocarcinoma within them
* No history of gastrointestinal cancer outside of the large bowel
* No other gastrointestinal mucosal epithelial disease (e.g., Barrett's esophagus, chronic or recurrent peptic ulcer disease, celiac sprue, or other disorders of nutrient absorption)
* No significant asymptomatic lesions on flexible sigmoidoscopy, such as inflammation, premalignancy or malignancy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* No platelet or coagulation abnormalities
* No personal or family history of a bleeding disorder
* Hematopoietic concentration must not be due to significant acute or chronic disorder

Hepatic:

* No liver disease

Renal:

* No renal insufficiency

Cardiovascular:

* No uncontrolled hypertension
* No chronic congestive heart failure
* No history of endocarditis
* No history of rheumatic fever
* No cardiac valve prostheses
* No mitral valve prolapse that requires antibiotic prophylaxis

Other:

* HIV negative
* No gout
* No pancreatitis
* No other chronic viral infection
* No significant acute or uncontrolled chronic medical illness
* Generally non-smoking (no more than 4 cigarettes per week, i.e., not daily smokers)
* Must abstain from smoking for at least 1 month prior to enrolling in the study
* No alcohol consumption of greater than 2 glasses of wine or beer per day
* Normal weight (90-120% of optimum body weight) and body habitus
* No change in weight within 5-10% of body weight within the past year
* No history of inflammatory bowel disease (either ulcerative colitis or Crohn's disease )
* No hearing or equilibrium disorders
* No other prior malignancy except resected carcinoma in situ of the cervix or nonmelanoma skin cancer
* No allergies to sulindac or tartrazine dyes or prior severe adverse reactions to nonsteroidal antiinflammatory drugs (asthma, gastrointestinal bleeding, or renal insufficiency)
* No potential allergy to curcumin, quercetin, or rutin
* No gastrointestinal bleeding
* Not institutionalized, mentally disabled, or incarcerated
* No unusually high intake of stored micronutrients or high doses of supplemental calcium or folate
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent coumadin
* No chronic use of nonsteroidal antiinflammatory drugs (unless they can be stopped for 3 months)
* No other putative colon cancer chemoprevention agents (unless they can be stopped for 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Shiff, MD, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rockefeller University Hospital, New York, New York, United States